CLINICAL TRIAL: NCT01672099
Title: The Effects of a Vitamin K-enriched Dairy Product on Vitamin K-status
Brief Title: Effects of Dairy on Vitamin K-status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-3-037
Record Dates: First submitted 2012-07-09; First posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Vitamin K-status; Vascular Health
Keywords: vitamin K2; menaquinone-7; vascular health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- nutrient enriched dairy (Active Comparator): Yoghurt product which contains vitamin K2 and extra dairy nutrients; all in a concentration of 15% of the recommended allowed daily intake (RDI)
  Interventions: Dietary Supplement: nutrient enriched product
- Basic dairy (Placebo Comparator): 2 basic yoghurt products
  Interventions: Dietary Supplement: basic dairy product

INTERVENTIONS:
Dietary Supplement: nutrient enriched product — The intervention in this study consists of the consumption of two nutrient enriched yoghurt products. The participants consume the study products twice a day during 12 weeks, one yoghurt product (250 ml) during breakfast and one yoghurt product (250 ml) during dinner.
  Arms: nutrient enriched dairy
Dietary Supplement: basic dairy product — The intervention in this study consists of the consumption of two basic yoghurt products. The participants consume the basic yoghurt products twice a day during 12 weeks, one yoghurt product (250 ml) during breakfast and one yoghurt product (250 ml) during dinner.
  Arms: Basic dairy

SUMMARY:
In this study, the beneficial effect of a nutrient enriched dairy product will be investigated on vitamin K-status. To achive this benefit, the study product contains extra vitamin K2. In addition, extra dairy minerals have been added to the study product that may support general health.

DETAILED DESCRIPTION:
In earlier studies, cardiovascular disease and osteoporosis were found to be associated with K2 intake, notably the higher menaquinones, MK-7, MK-8 and MK-9. Of these higher menaquinones, MK-7 was suggested to be the most effective form with respect to intestinal absorption, biologic half-life time, and efficacy on circulating biochemical markers. MK-7 is a natural product that is found in cheese, curd, and the Japanese food natto. Therefore, a nutrient enriched dairy product has been developed containing MK-7. The efficacy of this new product will be investigated on vitamin K status and on general health markers.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and postmenopausal women between 45 and 65 years old
* Subjects of body weight and height according to BMI between 23 and 30 kg/m2
* Subjects of Caucasian race
* Subject has given written consent to take part in the study
* Low vitamin K-status

Exclusion Criteria:

* Subjects with hypertension
* Subjects with hypercholesterolemia
* Subjects with (a history of) metabolic or gastrointestinal disease
* Subjects presenting chronic degenerative and/or inflammatory disease
* Subjects with (a history) of diabetes mellitus
* Abuse of drugs and/or alcohol
* Subjects receiving corticosteroϊd treatment
* Subjects using oral anticoagulants and subjects with clotting disorders
* Subjects using blood pressure lowering medication
* Subjects using cholesterol-lowering medication
* Subjects using multivitamins or vitamin K supplements
* Subjects consuming high amounts of vitamin K-containing food products
* Subjects with cow's milk allergy and lactose intolerance

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
undercarboxylated and carboxylated matrix-gla protein | 12 weeks
  The purpose of this study is to investigate the nutrient enriched product on vitamin K status as determined from the carboxylation status of Matrix Gla Protein

SECONDARY OUTCOMES:
undercarboxylated and carboxylated osteocalcin | 12 weeks
  The second purpose of this study is to investigate the nutrient enriched product on vitamin K status as determined from the carboxylation status of the vitamin K-dependent protein osteocalcin

OTHER OUTCOMES:
markers of vascular health and inflammation | 12 weeks
  The secondary purpose of this study is to investigate the nutrient enriched product on markers of vascular and general health

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — VitaK BV Maastricht University
Locations (1):
- Vitak BV / Maastricht University Medical Center, Maastricht, Netherlands